CLINICAL TRIAL: NCT04137224
Title: A Multicenter, Randomized, Open-label, Crossover, Phase 2 Study to Evaluate the Safety and Pharmacokinetics of IgPro20 (Subcutaneous Immunoglobulin, Hizentra®) and IgPro10 (Intravenous Immunoglobulin, Privigen®) in Adults With Systemic Sclerosis (SSc)
Brief Title: Safety and Pharmacokinetics of IgPro20 and IgPro10 in Adults With Systemic Sclerosis (SSc)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IgPro20_2001; 2018-003149-41 (EudraCT Number)
Record Dates: First submitted 2019-10-21; First posted 2019-10-23 (Actual); Results first posted 2024-02-05 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2023-05

CONDITIONS: Diffuse Cutaneous Systemic Sclerosis
Keywords: scleroderma
MeSH Terms: conditions — Scleroderma, Diffuse | interventions — Hizentra; Immunoglobulins, Intravenous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence A (IgPro20/IgPro10) (Experimental): Participants received IgPro20 of a total dose of 0.5 grams per kilogram (g/kg) over 2 sessions per week as a subcutaneous (SC) injection for up to 16 weeks in Treatment Period 1 followed by IgPro10 of a total dose of 2 g/kg over 2 to 5 sessions on consecutive days every 4 weeks as an intravenous (IV) infusion for up to 16 weeks in Treatment Period 2.
  Interventions: Biological: IgPro20; Biological: IgPro10
- Sequence B (IgPro10/IgPro20) (Experimental): Participants received IgPro10 of a total dose of 2 g/kg over 2 to 5 sessions on consecutive days every 4 weeks as an IV infusion for up to 16 weeks in Treatment Period 1 followed by IgPro20 of a total dose of 0.5 g/kg over 2 sessions per week as a SC injection for up to 16 weeks in Treatment Period 2.
  Interventions: Biological: IgPro20; Biological: IgPro10

INTERVENTIONS:
Biological: IgPro20 — Human normal immunoglobulin for subcutaneous administration
  Other Names: Hizentra
Biological: IgPro10 — Human normal immunoglobulin for intravenous administration
  Other Names: Privigen

SUMMARY:
This is a prospective, multicenter, randomized, open-label, crossover study to investigate the safety, tolerability, and pharmacokinetics of IgPro20 in participants with diffuse cutaneous systemic sclerosis (dcSSc). The pharmacokinetic study aims to evaluate the relative bioavailability of IgPro20, and characterize pharmacokinetics of IgPro20 and IgPro10, respectively, in participants with dcSSc. Safety, tolerability, and pharmacokinetics of IgPro10 will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years (male or female) at time of providing written informed consent
* Documented diagnosis of systemic sclerosis (scleroderma) according to American College of Rheumatology (ACR) and European League Against Rheumatism (EULAR) criteria 2013 (diffuse cutaneous form of SSc).
* Modified Rodnan Skin Score (mRSS) ≥ 15 and ≤ 45 at screening
* Disease duration ≤ 5 years defined as the time from the first non-Raynaud's phenomenon manifestation
* Capable of providing written informed consent and willing and able to adhere to all protocol requirements

Exclusion Criteria:

* Primary rheumatic autoimmune disease other than dcSSc, including but not limited to rheumatoid arthritis, systemic lupus erythematosus, mixed connective tissue disorder, polymyositis, dermatomyositis, as determined by the investigator. Note: Participants with fibromyalgia, secondary Sjogren's syndrome, and scleroderma-associated myopathy at screening are not excluded
* Participants has mRSS > 2 at the potential subcutaneous (SC) injection sites
* History of skin condition precluding SC infusion, or clinical signs and symptoms of a chronic skin disease other than systemic sclerosis or skin manifestation of an allergic disease or other dermatological conditions that would interfere with trial assessments or compromise safety (eg, dermatitis, eczema, psoriasis)
* Participants has clinical signs and symptoms of skin irritation (eg, pruritus, burning, erythema) or hypo/ hyperpigmentation (eg, scars, tattoos) at the potential SC injection sites
* Significant pulmonary arterial hypertension as documented by mean pulmonary arterial pressure > 30 mmHg on right heart catheterization requiring SC or IV prostacyclin or use of dual oral therapies
* Forced vital capacity < 50% predicted or a diffusing capacity of the lung for carbon dioxide (DLCO) ≤ 40% predicted (corrected for hemoglobin)
* A female who is pregnant, breastfeeding, or is a woman of childbearing potential who does not agree to use acceptable methods of contraception; a male who does agree to use acceptable methods of contraception.
* Evidence of chronic kidney disease with an estimated glomerular filtration rate (eGFR) < 45 mL/min/1.73m2 or if participants are receiving dialysis. Participants with current confirmed diagnosis of diabetes mellitus requiring medication with an eGFR < 90 ml/min/1.73m2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2019-09-19 (Actual); Primary Completion 2022-05-17 (Actual); Study Completion 2022-05-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — CSL Behring
Locations (9):
- Royal Adelaide Hospital, Adelaide, South Australia, Australia
- Germany (2):
  - Charité Universitätsmedizin Berlin, Berlin
  - Uniklinik Köln, innere Medizin, Cologne
- Italy (2):
  - ASST Spedali Civili di Brescia, Brescia
  - Azienda Ospedaliera Gaetano Pini, Milan
- Poland (3):
  - Uniwersytecki Szpital Kliniczny W Bialymstoku, Bialystok
  - Szpital Kliniczny Jezus, Warsaw
  - Narodowy Instytut Geriatrii, Warsaw
- The Royal Free Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
CSL will consider requests to share Individual Patient Data (IPD) from systematic review groups or bona-fide researchers. For information on the process and requirements for submitting a voluntary data sharing request for IPD, please contact CSL at clinicaltrials@cslbehring.com.
  Applicable country specific privacy and other laws and regulations will be considered and may prevent sharing of IPD.
  If the request is approved and the researcher has executed an appropriate data sharing agreement, IPD that has been appropriately anonymized will be available.
Supporting Information: Study Protocol, SAP
Time Frame: IPD requests may be submitted to CSL no earlier than 12 months after publication of the results of this study via an article made available on a public website.
Access Criteria: Requests may only be made by systematic review groups or bona-fide researchers whose proposed use of the IPD is non-commercial in nature and has been approved by an internal review committee.
  An IPD request will not be considered by CSL unless the proposed research question seeks to answer a significant and unknown medical science or patient care question as determined by CSL's internal review committee.
  The requesting party must execute an appropriate data sharing agreement before IPD will be made available.

REFERENCES:
- [Derived] Denton CP, Kowal-Bielecka O, Proudman SM, Olesinska M, Worm M, Del Papa N, Matucci-Cerinic M, Radewonuk J, Jochems J, Panaite A, Shebl A, Krupa A, Allanore Y, Hofmann JH, Gasior MJ. A phase 2 randomized trial of safety and pharmacokinetics of IgPro20 and IgPro10 in patients with diffuse cutaneous systemic sclerosis. Rheumatology (Oxford). 2025 Jun 1;64(6):3657-3666. doi: 10.1093/rheumatology/keaf066. PMID 39909490

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study centers in Australia, Germany, Italy, Poland, and the United Kingdom from 19 September 2019 to 17 May 2022.
Pre-assignment Details: A total of 30 participants were screened, of which 27 participants were enrolled and randomized to Sequence A or Sequence B in this study.
Period: Treatment Period 1 (Week 1 to Week 16)
Arm/Group | Sequence A (IgPro20/IgPro10) | Sequence B (IgPro10/IgPro20)
Started | 13 | 14
Completed | 12 | 13
Not Completed | 1 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1
Period: Treatment Period 2 (Week 17 to Week 32)
Arm/Group | Sequence A (IgPro20/IgPro10) | Sequence B (IgPro10/IgPro20)
Started | 13 (One participant who discontinued treatment period 1 due to Coronavirus disease (COVID) had entered treatment period 2.) | 13
Completed | 13 | 12
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants who received at least 1 infusion of IgPro20 or IgPro10.
Groups:
- Sequence A (IgPro20/IgPro10): Participants received IgPro20 of a total dose of 0.5 g/kg over 2 sessions per week as an SC injection for up to 16 weeks in Treatment Period 1 followed by IgPro10 of a total dose of 2 g/kg over 2 to 5 sessions on consecutive days every 4 weeks as an IV infusion for up to 16 weeks in Treatment Period 2.
- Total: Total of all reporting groups
Arm/Group | Sequence A (IgPro20/IgPro10) | Sequence B (IgPro10/IgPro20) | Total
Number analyzed (Participants) | 13 | 14 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.4 (12.22) | 47.4 (12.91) | 49.3 (12.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 8 | 18
  Male | 3 | 6 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 12 | 14 | 26
  Unknown or Not Reported | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 13 | 13 | 26
  Race: Other | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  Poland | 9 | 8 | 17
  United Kingdom | 3 | 3 | 6
  Italy | 1 | 0 | 1
  Australia | 0 | 2 | 2
  Germany | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With at Least One Adverse Event (AE) for IgPro20
Description: AE is any untoward medical occurrence in a patient or clinical investigation participant administered with a pharmaceutical product which does not necessarily have a causal relationship with the treatment. An AE can be any unfavorable and unintended sign (including an abnormal, clinically significant laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not considered related to the medicinal (investigational) product.
Time Frame: From first dose of study drug through last follow-up visit (up to 36 weeks)
Population: Safety analysis set included all participants who received at least 1 infusion of IgPro20 or IgPro10. Participants who received IgPro20 were analyzed.
Measure: Count of Participants; unit: Participants
Groups:
- Sequence A: IgPro20: Participants received IgPro20 of a total dose of 0.5 g/kg over 2 sessions per week as SC injection for up to 16 weeks in Treatment Period 1.
- Sequence B: IgPro20: Participants received IgPro20 of a total dose of 0.5 g/kg over 2 sessions per week as a SC injection for up to 16 weeks in Treatment Period 2.
Arm/Group | Sequence A: IgPro20 | Sequence B: IgPro20
Number analyzed (Participants) | 13 | 13
Participants | 9 | 9

2. Primary Outcome: Percentage of Participants With at Least One AE for IgPro20
Description: AE is any untoward medical occurrence in a patient or clinical investigation participant administered with a pharmaceutical product and which does not necessarily have a causal relationship with the treatment. An AE can be any unfavorable and unintended sign (including an abnormal, clinically significant laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not considered related to the medicinal (investigational) product.
Time Frame: From first dose of study drug through last follow-up visit (up to 36 weeks)
Population: Safety analysis set included all participants who received at least 1 infusion of IgPro20 or IgPro10. Participants who received IgPro20 were analyzed. The percentage of participants are rounded off to the single decimal point.
Measure: Number; unit: percentage of participants
Arm/Group | Sequence A: IgPro20 | Sequence B: IgPro20
Number analyzed (Participants) | 13 | 13
percentage of participants | 69.2 | 69.2

3. Primary Outcome: Number of Participants With at Least One Treatment-Emergent Adverse Event (TEAE) for IgPro20
Description: AE is any untoward medical occurrence in a patient or clinical investigation participant administered with a pharmaceutical product that does not necessarily have a causal relationship with the treatment. An AE can be any unfavorable and unintended sign (including an abnormal, clinically significant laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not considered related to the medicinal (investigational) product. TEAEs are defined as AEs reported at or after the start of the first infusion in the study.
Time Frame: From first dose of study drug through last follow-up visit (up to 36 weeks)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Sequence A: IgPro20 | Sequence B: IgPro20
Number analyzed (Participants) | 13 | 13
Participants | 9 | 9

4. Primary Outcome: Percentage of Participants With at Least One TEAE for IgPro20
Description: AE is any untoward medical occurrence in a patient or clinical investigation participant administered with a pharmaceutical product and which does not necessarily have a causal relationship with the treatment. An AE can be any unfavorable and unintended sign (including an abnormal, clinically significant laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not considered related to the medicinal (investigational) product. TEAEs are defined as AEs reported at or after the start of the first infusion in the study.
Time Frame: From first dose of study drug through last follow-up visit (up to 36 weeks)
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Sequence A: IgPro20 | Sequence B: IgPro20
Number analyzed (Participants) | 13 | 13
percentage of participants | 69.2 | 69.2

5. Primary Outcome: Number of Participants With at Least One Serious Adverse Event (SAE) for IgPro20
Description: An SAE is defined as any untoward medical occurrence that at any dose results in death, is life-threatening, requires in-patient hospitalization or prolongation of existing hospitalization, is a congenital anomaly or birth defect, or is a medically significant event.
Time Frame: From first dose of study drug through last follow-up visit (up to 36 weeks)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Sequence A: IgPro20 | Sequence B: IgPro20
Number analyzed (Participants) | 13 | 13
Participants | 2 | 3

6. Primary Outcome: Percentage of Participants With at Least One SAE for IgPro20
Description: as for outcome 5
Time Frame: From first dose of study drug through last follow-up visit (up to 36 weeks)
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Groups:
- Sequence A: IgPro20: Participants received IgPro20 of a total dose of 0.5 g/kg over 2 sessions per week as a SC injection for up to 16 weeks in Treatment Period 1.
Arm/Group | Sequence A: IgPro20 | Sequence B: IgPro20
Number analyzed (Participants) | 13 | 13
percentage of participants | 15.4 | 23.1

7. Primary Outcome: Number of Participants With at Least One Adverse Event of Special Interest (AESI) for IgPro20
Description: AE is any untoward medical occurrence in a patient or clinical investigation participant administered with a pharmaceutical product and which does not necessarily have a causal relationship with the treatment. An AE can be any unfavorable and unintended sign (including an abnormal, clinically significant laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not considered related to the medicinal (investigational) product. An AESI is an AE of scientific and medical concern specific to the sponsor's product or program, for which ongoing monitoring and rapid communication by the investigator to the sponsor is appropriate.
Time Frame: From first dose of study drug through last follow-up visit (up to 36 weeks)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Sequence A: IgPro20 | Sequence B: IgPro20
Number analyzed (Participants) | 13 | 13
Participants | 0 | 1

8. Primary Outcome: Percentage of Participants With at Least One AESI for IgPro20
Description: as for outcome 7
Time Frame: From first dose of study drug through last follow up visit (up to 36 weeks)
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Sequence A: IgPro20 | Sequence B: IgPro20
Number analyzed (Participants) | 13 | 13
percentage of participants | 0 | 7.7

9. Primary Outcome: Number of Participants With AEs Categorized as Infusion Site Reactions (ISRs) for IgPro20
Description: ISRs included all events reported within the MedDRA high-level terms 'Administration site reactions', 'Infusion site reactions', or 'Injection site reactions'.
Time Frame: From first dose of study drug through last follow up visit (up to 36 weeks)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Sequence A: IgPro20 | Sequence B: IgPro20
Number analyzed (Participants) | 13 | 13
Participants | 2 | 3

10. Primary Outcome: Percentage of Participants With AEs Categorized as ISRs for IgPro20
Description: as for outcome 9
Time Frame: From first dose of study drug through last follow up visit (up to 36 weeks)
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Sequence A: IgPro20 | Sequence B: IgPro20
Number analyzed (Participants) | 13 | 13
percentage of participants | 15.4 | 23.1

11. Primary Outcome: Rate of ISRs Per Infusion for IgPro20
Description: ISR rate per infusion = total number of ISRs across all participants while on IgPro20 / total number of IgPro20 Infusions across all participants. ISRs included all events reported within the MedDRA high-level terms 'Administration site reactions NEC', 'Infusion site reactions', or 'Injection site reactions'
Time Frame: From first dose of study drug through last follow up visit (up to 36 weeks)
Population: as for outcome 1
Measure: Number; unit: ISRs per infusion
Units Other Than Participants: Infusions
Arm/Group | Sequence A: IgPro20 | Sequence B: IgPro20
Number analyzed (Participants) | 13 | 13
Number analyzed (Infusions) | 353 | 333
ISRs per infusion | 0.0057 | 0.0360

12. Primary Outcome: Time to Onset of ISRs for IgPro20
Description: ISRs included all events reported within the MedDRA high-level terms 'Administration site reactions', 'Infusion site reactions', or 'Injection site reactions'. Time to onset of ISR since the start of the treatment period was reported.
Time Frame: From first dose of study drug through last follow up visit (up to 36 weeks)
Population: Safety analysis set included all participants who received at least 1 infusion of IgPro20 or IgPro10. Participants who received IgPro20 and with ISRs were analyzed.
Measure: Median (Full Range); unit: days
Units Other Than Participants: ISRs
Arm/Group | Sequence A: IgPro20 | Sequence B: IgPro20
Number analyzed (Participants) | 2 | 3
Number analyzed (ISRs) | 2 | 12
days | 2.0 [1 to 3] | 15.0 [1 to 64]

13. Primary Outcome: Duration of ISRs for IgPro20
Description: as for outcome 9
Time Frame: From first dose of study drug through last follow up visit (up to 36 weeks)
Population: as for outcome 12
Measure: Median (Full Range); unit: minutes
Units Other Than Participants: ISRs
Arm/Group | Sequence A: IgPro20 | Sequence B: IgPro20
Number analyzed (Participants) | 2 | 3
Number analyzed (ISRs) | 2 | 12
minutes | 162.0 [162 to 162] | 220.0 [180 to 1170]

14. Primary Outcome: Number of Participants With Clinically Significant Abnormalities in Laboratory Tests for IgPro20
Description: Abnormality criteria:Hematology-Hemoglobin:<10 g/dL;Platelet count:<75x10^9/L or >500x10^9/L;White Blood Cell Count:<3x10^9/L or >16x10^9/L;Neutrophils:absolute <1.5x10^9/L,differential <40%;Lymphocytes:absolute <0.8x10^9/L,differential <10 or >50%; Biochemistry-Bilirubin:>1.5xupper limit of normal (ULN);Alkaline phosphatase:>2.5xULN;Serum Glutamic-oxalacetic transaminase(SGOT), Aspartate transaminase(AST):>3xULN;Serum glutamic-pyruvic transaminase(SGPT), Alanine transaminase(ALT):>3xULN;Screening:AST/ALT >3xULN and Total Bilirubin >2xULN;Urea nitrogen:>2.5xULN; Creatinine, serum>1.5xbaseline assessment or change >0.3mg/dL since last visit;Glucose,blood (non-fasting):<55/>160mg/dL;Calcium:<7/>11.5mg/dL;Total protein: <5/>9g/dL; Albumin:<3g/dL;Sodium:<130/>150mmol/L;Potassium:<3/>5.5mmol/L; Uric acid,serum:>10mg/dL Males,>8mg/dL Females;Gamma Glutamyl Transpeptidase:>2.5xULN; Phosphorus,inorganic:<2.5/>5mg/dL;Lactate dehydrogenase:>3xULN;Urinalysis-Protein:>20mg/dL.
Time Frame: From first dose of study drug through last follow up visit (up to 36 weeks)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Sequence A: IgPro20 | Sequence B: IgPro20
Number analyzed (Participants) | 13 | 13
Participants | 0 | 0

15. Primary Outcome: Number of Participants With Clinically Significant Changes in Vital Signs for IgPro20
Description: Clinically significant abnormality criteria for vital signs included Systolic blood pressure (BP): <100 millimeters of mercury (mmHg) or ≥140 mmHg or ≥140 mmHg and increase >10 from reference visit; Diastolic BP: <50 mmHg or ≥90 mmHg or ≥90 mmHg and increase >10 from reference visit; Pulse rate: <50 beats/minute or ≥120 beats/minute or ≥120 beats/minute and increase >15 from reference visit; Weight (kilograms) ≥10% change (increase and decrease) from baseline assessment; Body temperature: > 39-degree Celsius (°C ) or <35°C (oral, tympanic, axilla or forehead).
Time Frame: From first dose of study drug through last follow up visit (up to 36 weeks)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Sequence A: IgPro20 | Sequence B: IgPro20
Number analyzed (Participants) | 13 | 13
Participants | 0 | 0

16. Primary Outcome: Number of Participants With Clinically Significant Abnormalities in Electrocardiogram (ECG) Parameters for IgPro20
Description: Clinically significant abnormality criteria for ECG parameters included Heart rate: ≤50 or ≥100 beats/minute; PR Interval: ≥200 millisecond (msec); QRS Interval: ≥120 msec; QT: ≥480 msec; QT interval corrected using Bazett' s formula (QTcB): ≤ 500 msec; QT interval corrected using Fridericia's formula (QTcF): >500 msec; QT: increase from baseline ≥ 30; QTcB: increase from baseline < 60 msec; QTcF: increase from baseline ≥ 60.
Time Frame: From first dose of study drug through last follow up visit (up to 36 weeks)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Sequence A: IgPro20 | Sequence B: IgPro20
Number analyzed (Participants) | 13 | 13
Participants | 0 | 1

17. Primary Outcome: Number of Participants With Clinically Significant Abnormalities in Pulmonary Function Tests (PFTs) for IgPro20
Description: PFTs include Spirometry which included forced vital capacity (FVC) % Predicted, considered as clinically significant abnormality when decrease is greater than10 percentage points from the reference visit.
Time Frame: From first dose of study drug through last follow up visit (up to 36 weeks)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Sequence A: IgPro20 | Sequence B: IgPro20
Number analyzed (Participants) | 13 | 13
Participants | 0 | 0

18. Secondary Outcome: Relative Bioavailability (%F) of IgPro20
Description: Relative bioavailability was calculated using Mixed Model Repeated Measures on Log-transformed Dose-normalized area under the curve to the end of the dosing period [AUC0-tau] following administration of the first dose of IgPro20 in the last week of dosing for Sequence A and / or Sequence B. Relative Bioavailability= (AUCtau IgPro20 (SC)/dose of IgPro20 (SC) / (AUCtau of IgPro10 (IV)/dose of IgPro10 (IV)).
Time Frame: Seq A-(Pre-injection [inj] at Weeks [Wks] 1,5,9,13,14; 24,48,72,96,168 hours [hrs] post 1st inj at Wk 14; 240 hrs post 1st inj at Wk 15), Seq B-(Pre-inj at Wks 17,21,25,29,30; 24,48,72,96,168 hrs post 1st inj at Wk 30; 240 hrs post 1st inj at Wk 31)
Population: Safety analysis set included all participants who received at least 1 infusion of IgPro20 or IgPro10. 'Overall number of participants analyzed' indicates the number of participants who received IgPro20 and with data available for outcome measure analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: percentage bioavailability
Arm/Group | Sequence A: IgPro20 | Sequence B: IgPro20
Number analyzed (Participants) | 12 | 12
percentage bioavailability | 0.831 [0.7343 to 0.9396] | 0.698 [0.6235 to 0.7804]

19. Secondary Outcome: Area Under the Concentration Curve to the End of the Dosing Period (AUC0-tau) for IgPro20
Time Frame: as for outcome 18
Population: as for outcome 18
Measure: Geometric Mean (95% Confidence Interval); unit: hours*grams per liter (h*g/L)
Arm/Group | Sequence A: IgPro20 | Sequence B: IgPro20
Number analyzed (Participants) | 12 | 11
hours*grams per liter (h*g/L) | 3835.68 [3394.749 to 4333.883] | 3581.08 [3326.635 to 3854.997]

20. Secondary Outcome: Area Under the Concentration Curve up to the Last Measurable Concentration (AUC0-last) for IgPro20
Time Frame: as for outcome 18
Population: as for outcome 18
Measure: Geometric Mean (95% Confidence Interval); unit: h*g/L
Arm/Group | Sequence A: IgPro20 | Sequence B: IgPro20
Number analyzed (Participants) | 12 | 12
h*g/L | 5361.61 [4729.962 to 6077.619] | 4898.02 [4437.732 to 5406.046]

21. Secondary Outcome: Maximum Plasma Drug Concentration (Cmax) for IgPro20
Time Frame: as for outcome 18
Population: as for outcome 18
Measure: Geometric Mean (95% Confidence Interval); unit: g/L
Arm/Group | Sequence A: IgPro20 | Sequence B: IgPro20
Number analyzed (Participants) | 12 | 12
g/L | 24.237 [21.6041 to 27.1898] | 23.203 [21.7278 to 24.7782]

22. Secondary Outcome: Minimum Plasma Drug Concentration (Ctrough) for IgPro20 in Sequence A
Time Frame: Pre-injection at Weeks 5, 9, 13, and 14
Population: Safety analysis set included all participants who received at least 1 infusion of IgPro20 or IgPro10. Participants who received IgPro20 were analyzed. 'Number analyzed' indicates the number of participants with data available for analysis at the specified time point.
Measure: Geometric Mean (Full Range); unit: g/L
Arm/Group | Sequence A: IgPro20
Number analyzed (Participants) | 13
g/L
  Week 5: number analyzed (Participants) | 12
  Week 5 | 22.046 [16.69 to 63.70]
  Week 9 | 21.950 [14.71 to 30.51]
  Week 13: number analyzed (Participants) | 12
  Week 13 | 22.354 [16.98 to 31.36]
  Week 14: number analyzed (Participants) | 12
  Week 14 | 21.814 [14.49 to 27.93]

23. Secondary Outcome: Minimum Plasma Drug Concentration (Ctrough) for IgPro20 in Sequence B
Time Frame: Pre-injection at Weeks 21, 25, 29, and 30
Population: as for outcome 18
Measure: Geometric Mean (Full Range); unit: g/L
Arm/Group | Sequence B: IgPro20
Number analyzed (Participants) | 12
g/L
  Week 21 | 20.427 [12.82 to 25.48]
  Week 25 | 21.603 [16.92 to 30.49]
  Week 29 | 21.903 [18.89 to 28.47]
  Week 30 | 20.497 [18.15 to 23.59]

24. Secondary Outcome: Area Under the Concentration Curve to the End of the Dosing Period (AUC0-tau) for IgPro10
Time Frame: Seq A and B respectively-Pre-infusion (inf) at Wks 17,21,25,29 and 1,5,9,13; 1 hour (hr) post 1st and 2nd inf, 168 hr post 1st inf at Wk 29,13; 264 and 336 hr post 1st inf at Wk 30, 14; 504 hr post 1st inf at Wk 31,15; 672 hr post 1st inf at Wk 32,16
Population: Safety analysis set included all participants who received at least 1 infusion of IgPro20 or IgPro10. 'Overall number of participants analyzed' indicates the number of participants who received IgPro10 and with data available for outcome measure analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: h*g/L
Groups:
- Sequence A: IgPro10: Participants received IgPro10 of a total dose of 2 g/kg over 2 to 5 sessions on consecutive days every 4 weeks as an IV infusion for up to 16 weeks in Treatment Period 2.
- Sequence B: IgPro10: Participants received IgPro10 of a total dose of 2 g/kg over 2 to 5 sessions on consecutive days every 4 weeks as an IV infusion for up to 16 weeks in Treatment Period 1.
Arm/Group | Sequence A: IgPro10 | Sequence B: IgPro10
Number analyzed (Participants) | 12 | 12
h*g/L | 16942.66 [15097.493 to 19013.345] | 17672.03 [16402.479 to 19039.837]

25. Secondary Outcome: Area Under the Concentration Curve up to the Last Measurable Concentration (AUC0-last) for IgPro10
Time Frame: as for outcome 24
Population: as for outcome 24
Measure: Geometric Mean (95% Confidence Interval); unit: h*g/L
Arm/Group | Sequence A: IgPro10 | Sequence B: IgPro10
Number analyzed (Participants) | 13 | 12
h*g/L | 16520.48 [14742.232 to 18513.218] | 17349.72 [15917.101 to 18911.275]

26. Secondary Outcome: Maximum Plasma Drug Concentration (Cmax) for IgPro10
Time Frame: as for outcome 24
Population: as for outcome 24
Measure: Geometric Mean (95% Confidence Interval); unit: g/L
Arm/Group | Sequence A: IgPro10 | Sequence B: IgPro10
Number analyzed (Participants) | 13 | 12
g/L | 47.142 [41.2538 to 53.8713] | 44.996 [39.2110 to 51.6340]

27. Secondary Outcome: Minimum Plasma Drug Concentration (Ctrough) for IgPro10 in Sequence A
Time Frame: Pre-infusion at Weeks 21, 25 and 29
Population: Safety analysis set included all participants who received at least 1 infusion of IgPro20 or IgPro10. Participants who received IgPro10 were analyzed. 'Number analyzed' indicates the number of participants with data available for analysis at the specified time point.
Measure: Geometric Mean (Full Range); unit: g/L
Groups:
- Sequence A: IgPro10: Participants received IgPro10 of a total dose of 2g/kg over 2 to 5 sessions on consecutive days every 4 weeks as an IV infusion for up to 16 weeks in Treatment Period 2.
Arm/Group | Sequence A: IgPro10
Number analyzed (Participants) | 13
g/L
  Week 21: number analyzed (Participants) | 12
  Week 21 | 16.123 [9.69 to 34.70]
  Week 25 | 17.497 [8.80 to 54.96]
  Week 29 | 16.838 [8.51 to 58.16]

28. Secondary Outcome: Minimum Plasma Drug Concentration (Ctrough) for IgPro10 in Sequence B
Time Frame: Pre-infusion at Weeks 5, 9 and 13
Population: Safety analysis set included all participants who received at least 1 infusion of IgPro20 or IgPro10. 'Overall number of participants analyzed' indicates the number of participants who received IgPro10 and with data available for outcome measure analysis. 'Number analyzed' indicates the number of participants with data available for analysis at the specified time point.
Measure: Geometric Mean (Full Range); unit: g/L
Arm/Group | Sequence B: IgPro10
Number analyzed (Participants) | 13
g/L
  Week 5: number analyzed (Participants) | 12
  Week 5 | 17.104 [12.77 to 24.04]
  Week 9 | 17.744 [13.92 to 23.36]
  Week 13 | 17.113 [12.89 to 25.43]

29. Secondary Outcome: Number of Participants With at Least One AE for IgPro10
Description: as for outcome 1
Time Frame: From first dose of study drug through last follow up visit (up to 36 weeks)
Population: Safety analysis set included all participants who received at least 1 infusion of IgPro20 or IgPro10. Participants who received IgPro10 were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Sequence A: IgPro10 | Sequence B: IgPro10
Number analyzed (Participants) | 13 | 14
Participants | 5 | 8

30. Secondary Outcome: Percentage of Participants With at Least One AE for IgPro10
Description: as for outcome 1
Time Frame: From first dose of study drug through last follow up visit (up to 36 weeks)
Population: Safety analysis set included all participants who received at least 1 infusion of IgPro20 or IgPro10. Participants who received IgPro10 were analyzed. The percentage of participants are rounded off to the single decimal point.
Measure: Number; unit: percentage of participants
Arm/Group | Sequence A: IgPro10 | Sequence B: IgPro10
Number analyzed (Participants) | 13 | 14
percentage of participants | 38.5 | 57.1

31. Secondary Outcome: Number of Participants With at Least One TEAE for IgPro10
Description: as for outcome 3
Time Frame: From first dose of study drug through last follow up visit (up to 36 weeks)
Population: as for outcome 29
Measure: Count of Participants; unit: Participants
Arm/Group | Sequence A: IgPro10 | Sequence B: IgPro10
Number analyzed (Participants) | 13 | 14
Participants | 5 | 8

32. Secondary Outcome: Percentage of Participants With at Least One TEAE for IgPro10
Description: AE is any untoward medical occurrence in a patient or clinical investigation participant administered with a pharmaceutical product which does not necessarily have a causal relationship with the treatment. An AE can be any unfavorable and unintended sign (including an abnormal, clinically significant laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not considered related to the medicinal (investigational) product. TEAEs are defined as AEs reported at or after the start of the first infusion in the study.
Time Frame: From first dose of study drug through last follow up visit (up to 36 weeks)
Population: as for outcome 30
Measure: Number; unit: percentage of participants
Arm/Group | Sequence A: IgPro10 | Sequence B: IgPro10
Number analyzed (Participants) | 13 | 14
percentage of participants | 38.5 | 57.1

33. Secondary Outcome: Number of Participants With at Least One SAE for IgPro10
Description: as for outcome 5
Time Frame: From first dose of study drug through last follow up visit (up to 36 weeks)
Population: as for outcome 29
Measure: Count of Participants; unit: Participants
Arm/Group | Sequence A: IgPro10 | Sequence B: IgPro10
Number analyzed (Participants) | 13 | 14
Participants | 1 | 1

34. Secondary Outcome: Percentage of Participants With at Least One SAE for IgPro10
Description: as for outcome 5
Time Frame: From first dose of study drug through last follow up visit (up to 36 weeks)
Population: as for outcome 30
Measure: Number; unit: percentage of participants
Arm/Group | Sequence A: IgPro10 | Sequence B: IgPro10
Number analyzed (Participants) | 13 | 14
percentage of participants | 7.7 | 7.1

35. Secondary Outcome: Number of Participants With at Least One AESI for IgPro10
Description: as for outcome 7
Time Frame: From first dose of study drug through last follow up visit (up to 36 weeks)
Population: as for outcome 29
Measure: Count of Participants; unit: Participants
Arm/Group | Sequence A: IgPro10 | Sequence B: IgPro10
Number analyzed (Participants) | 13 | 14
Participants | 0 | 0

36. Secondary Outcome: Percentage of Participants With at Least One AESI for IgPro10
Description: as for outcome 7
Time Frame: From first dose of study drug through last follow up visit (up to 36 weeks)
Population: as for outcome 30
Measure: Number; unit: percentage of participants
Arm/Group | Sequence A: IgPro10 | Sequence B: IgPro10
Number analyzed (Participants) | 13 | 14
percentage of participants | 0 | 0

37. Secondary Outcome: Number of Participants With AEs Categorized as ISRs for IgPro10
Description: as for outcome 9
Time Frame: From first dose of study drug through last follow up visit (up to 36 weeks)
Population: as for outcome 29
Measure: Count of Participants; unit: Participants
Arm/Group | Sequence A: IgPro10 | Sequence B: IgPro10
Number analyzed (Participants) | 13 | 14
Participants | 0 | 0

38. Secondary Outcome: Percentage of Participants With AEs Categorized as ISRs for IgPro10
Description: as for outcome 9
Time Frame: From first dose of study drug through last follow up visit (up to 36 weeks)
Population: as for outcome 29
Measure: Number; unit: percentage of participants
Arm/Group | Sequence A: IgPro10 | Sequence B: IgPro10
Number analyzed (Participants) | 13 | 14
percentage of participants | 0 | 0

39. Secondary Outcome: Number of Participants With Clinically Significant Abnormalities in Laboratory Tests for IgPro10
Description: as for outcome 14
Time Frame: From first dose of study drug through last follow up visit (up to 36 weeks)
Population: as for outcome 29
Measure: Count of Participants; unit: Participants
Arm/Group | Sequence A: IgPro10 | Sequence B: IgPro10
Number analyzed (Participants) | 13 | 14
Participants | 0 | 0

40. Secondary Outcome: Number of Participants With Clinically Significant Changes in Vital Signs for IgPro10
Description: as for outcome 15
Time Frame: From first dose of study drug through last follow up visit (up to 36 weeks)
Population: as for outcome 29
Measure: Count of Participants; unit: Participants
Arm/Group | Sequence A: IgPro10 | Sequence B: IgPro10
Number analyzed (Participants) | 13 | 14
Participants | 0 | 0

41. Secondary Outcome: Number of Participants With Clinically Significant Abnormalities in ECG Parameters for IgPro10
Description: as for outcome 16
Time Frame: From first dose of study drug through last follow up visit (up to 36 weeks)
Population: as for outcome 29
Measure: Count of Participants; unit: Participants
Arm/Group | Sequence A: IgPro10 | Sequence B: IgPro10
Number analyzed (Participants) | 13 | 14
Participants | 0 | 0

42. Secondary Outcome: Number of Participants With Clinically Significant Abnormalities in PFTs for IgPro10
Description: as for outcome 17
Time Frame: From first dose of study drug through last follow up visit (up to 36 weeks)
Population: as for outcome 29
Measure: Count of Participants; unit: Participants
Arm/Group | Sequence A: IgPro10 | Sequence B: IgPro10
Number analyzed (Participants) | 13 | 14
Participants | 0 | 0

43. Other Pre Specified Outcome: Rate of ISRs Per Participant for IgPro20
Time Frame: From first dose of study drug through last follow up visit (up to 36 weeks)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From first dose of study drug through last follow up visit (up to 36 weeks)
Description: Safety analysis set included all participants who received at least 1 infusion of IgPro20 or IgPro10.
Arm/Group | Sequence A: IgPro20 | Sequence A: IgPro10 | Sequence B: IgPro10 | Sequence B: IgPro20
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13 | 0/14 | 0/13
Serious Adverse Events (participants affected / at risk) | 2/13 | 1/13 | 1/14 | 3/13
Other Adverse Events (participants affected / at risk) | 8/13 | 5/13 | 8/14 | 6/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sequence A: IgPro20 (N=13) | Sequence A: IgPro10 (N=13) | Sequence B: IgPro10 (N=14) | Sequence B: IgPro20 (N=13)
Viral Infection (Infections and infestations) | 0 | 0 | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 0 | 0
Chronic gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sequence A: IgPro20 (N=13) | Sequence A: IgPro10 (N=13) | Sequence B: IgPro10 (N=14) | Sequence B: IgPro20 (N=13)
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 2 | 1
Toothache (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Eructation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Saliva altered (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 5 | 0
Anosmia (Nervous system disorders) | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 1
Sciatica (Nervous system disorders) | 1 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 1 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Dermatitis psoriasiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Lichenoid keratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Scleroderma associated digital ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Umbilical erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Infusion site pain (General disorders) | 1 | 0 | 0 | 1
Infusion site swelling (General disorders) | 0 | 0 | 0 | 2
Fatigue (General disorders) | 0 | 0 | 0 | 1
Infusion site discharge (General disorders) | 0 | 0 | 0 | 1
Infusion site erosion (General disorders) | 0 | 0 | 0 | 1
Infusion site erythema (General disorders) | 0 | 0 | 0 | 1
Infusion site haemorrhage (General disorders) | 0 | 0 | 0 | 1
Infusion site reaction (General disorders) | 0 | 0 | 0 | 1
Infusion site vesicles (General disorders) | 0 | 0 | 0 | 1
Injection site hypersensitivity (General disorders) | 1 | 0 | 0 | 0
Injection site mass (General disorders) | 0 | 0 | 0 | 1
Peripheral swelling (General disorders) | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 0
COVID-19 (Infections and infestations) | 1 | 0 | 0 | 2
Gingivitis (Infections and infestations) | 0 | 0 | 1 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Dry eye (Eye disorders) | 1 | 0 | 0 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Depressed mood (Psychiatric disorders) | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2021-02-22): https://cdn.clinicaltrials.gov/large-docs/24/NCT04137224/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-09): https://cdn.clinicaltrials.gov/large-docs/24/NCT04137224/SAP_001.pdf